CLINICAL TRIAL: NCT00142909
Title: Lofexidine: Enhancing Naltrexone Treatment for Opiate Addiction
Brief Title: Effectiveness of Lofexidine to Prevent Stress-Related Opiate Relapse During Naltrexone Treatment - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Rajita Sinha, Professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-18219-1; R01-18219-1; DPMC
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Results first posted 2013-11-20 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Opioid-Related Disorders
Keywords: Opioid dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — lofexidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug: Lofexidine (Experimental): Lofexidine: Study medication
  Participants will receive daily lofexidine and the dosing will be initiated at 0.4 mg bid and increased to 0.8mg in week 1 and 1.0 and 1.2 mg bid in week 2, and maintained at 1.2mg bid for weeks 3 to 12. They are then tapered down to 0 over the course of four days in week 12. While the target dose will be 2.4 mg daily, if any subject shows reduced tolerability at this or a lower dose, the dose will be adjusted to the maximum tolerated dose for that subject.
  Interventions: Drug: Lofexidine
- Drug: Placebo (Placebo Comparator): Placebo pill.
  Participants will receive daily placebo and will follow the same scheduled delivery as those in the intervention for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lofexidine — Participants will receive lofexidine. The dosing will be initiation at 0.4 mg bid and increased to 0.8mg in week 1 and 1.0 and 1.2 mg bid in week 2, and maintained at 1.2mg bid for weeks 3 to 12. They are then tapered down to 0 over the course of four days in week 12. While the target dose will be 2.4 mg daily, if any subject shows reduced tolerability at this or a lower dose, the dose will be adjusted to the maximum tolerated dose for that subject.
  Arms: Drug: Lofexidine
Drug: Placebo — Lofexidine Placebo
  Arms: Drug: Placebo

SUMMARY:
Lofexidine is an experimental medication that may be beneficial in reducing opiate withdrawal symptoms, such as sleep difficulty, anxiety, and tension. The purpose of this study is to determine whether lofexidine in combination with naltrexone can improve an individual's ability to cope with stress and subsequently increase the chances of remaining abstinent from opiates.

DETAILED DESCRIPTION:
Naltrexone is a medication currently used to treat opiate dependence. Naltrexone blocks the euphoric effects of opiates. However, naltrexone treatment suffers from high rates of drop-out and relapse. One possible explanation for this is that opiate addicts continue to experience stress in early recovery from opiate dependence. Lofexidine is an experimental medication currently used in the United Kingdom for opiate detoxification and to treat opiate withdrawal symptoms, including sleep difficulty, muscle pain, anxiety, and tension. The purpose of this study is to examine whether lofexidine in combination with naltrexone can improve an individual's ability to cope with stress. The study will examine whether this, in turn, increases the likelihood that an individual remains abstinent from opiates and maintains recovery for a longer time period.

Participants in this 12-week, double-blind, placebo-controlled trial will be randomly assigned to receive either lofexidine or placebo while currently receiving standard naltrexone outpatient treatment. Lofexidine will be initiated at twice daily doses of 0.4 mg and increased to 0.8 mg by the end of Week 1. The doses will be increased to 1.2 mg by the end of Week 2, and maintained at this level for Weeks 3 through 12. During Week 12, lofexidine discontinuation will be tapered over 4 days. Hour-long study visits will occur 3 times each week to assess vital signs, medication side effects, and withdrawal symptoms. Blood, alcohol, and urine tests will be performed as well as a psychiatric evaluation. Administration of naltrexone will also occur 3 times each week. Follow-up visits will occur at Months 1 and 3 after discontinuation of lofexidine.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for opioid dependence
* Eligible to take a daily dose of 50 mg of naltrexone
* Normal EKG
* Able to read English

Exclusion Criteria:

* Currently psychotic or psychiatrically disabled (e.g., suicidal, homicidal, manic)
* Regular use of anticonvulsants, sedatives/hypnotics, prescription analgesics, antihypertensives (including clonidine), antiarrhythmics, antiretroviral medications, or tricyclic antidepressants
* Underlying medical conditions, such as cerebral, kidney, thyroid, or cardiac pathology, and currently taking medications for any of these conditions
* Abstinent from opiates for more than 4 weeks prior to initiation of naltrexone
* Medical problems precluding naltrexone treatment, such as hepato-cellular injury, as evidenced by abnormal liver enzyme tests (greater than three times the normal level) and a history of cirrhosis
* Hypotensive (resting blood pressure below 90/50 mm Hg)
* Pregnant or breastfeeding
* Use of an investigational drug within the 3 months prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2005-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajita Sinha, Principal Investigator — Yale University
Locations (1):
- Yale University, Psychiatry, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Lofexidine: Lofexidine: Study medication
  Participants will receive daily lofexidine and the dosing will be initiated at 0.4 mg bid and increased to 0.8mg in week 1 and 1.0 and 1.2 mg bid in week 2, and maintained at 1.2mg bid for weeks 3 to 12. They are then tapered down to 0 over the course of four days in week 12. While the target dose will be 2.4 mg daily, if any subject shows reduced tolerability at this or a lower dose, the dose will be adjusted to the maximum tolerated dose for that subject.
- Placebo: Participants will receive daily placebo and follow the same schedule as the active intervention for 12 weeks.
Period: Randomization
Arm/Group | Lofexidine | Placebo
Started | 42 | 44
Completed | 35 | 34
Not Completed | 7 | 10
Not completed — Various Reasons | 7 | 10
Period: Medications Begin
Arm/Group | Lofexidine | Placebo
Started | 35 | 34
Completed | 26 | 31
Not Completed | 9 | 3
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lofexidine | Placebo | Total
Number analyzed (Participants) | 35 | 34 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.63 (9.99) | 25.56 (7.66) | 26.24 (7.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 27 | 27 | 54
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 2 | 1 | 3
  Caucasian | 32 | 31 | 63
  Hispanic | 1 | 1 | 2
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: SOWS: the Subjective Opiate Withdrawal Scale
Description: The Subjective Opiate Withdrawal Scale (SOWS) consists of 16 symptoms rated in intensity by patients on a 5-point scale of intensity as follows: 0=not at all, 1=a little, 2=moderately, 3=quite a bit, 4=extremely. The total score is a sum of item ratings, and ranges from 0 to 64. The greater the score, the greater the intensity of Opiate Withdrawal. Source: Reprinted from Handelsman et al. 1987, p. 296, by courtesy of Marcel Dekker, Inc.Other Sources: Gossop 1990; Bradley et al. 1987. ACCESSED: http://www.ncbi.nlm.nih.gov/books/NBK64244/
Time Frame: 1 Week
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Lofexidine: Lofexidine: Study medication
- Placebo: Placebo pill
Arm/Group | Lofexidine | Placebo
Number analyzed (Participants) | 26 | 31
units on a scale | 11.5 (9.7) | 12.5 (6.7)

2. Secondary Outcome: Systolic Blood Pressure
Time Frame: 1 Week
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Lofexidine | Placebo
Number analyzed (Participants) | 26 | 31
mm Hg | 115.3 (10.1) | 126.0 (12.0)

3. Primary Outcome: SOWS: the Subjective Opiate Withdrawal Scale
Description: as for outcome 1
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lofexidine | Placebo
Number analyzed (Participants) | 26 | 31
units on a scale | 2.9 (5.8) | 5.0 (13.3)

4. Secondary Outcome: Systolic Blood Pressure
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Lofexidine | Placebo
Number analyzed (Participants) | 26 | 31
mm Hg | 122.3 (10.1) | 126.7 (8.9)

5. Secondary Outcome: Diastolic Blood Pressure
Time Frame: 1 Week
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Lofexidine | Placebo
Number analyzed (Participants) | 26 | 31
mm Hg | 68.2 (7.6) | 73.4 (7.6)

6. Secondary Outcome: Diastolic Blood Pressure
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Lofexidine | Placebo
Number analyzed (Participants) | 26 | 31
mm Hg | 74.4 (12.5) | 76.1 (7.8)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Lofexidine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/31
Other Adverse Events (participants affected / at risk) | 16/26 | 14/31
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lofexidine (N=26) | Placebo (N=31)
Headache (Nervous system disorders) | 9 (9) | 10 (10)
Dizzy/lightheaded (Nervous system disorders) | 9 (9) | 3 (3)
Tired/fatigued (Nervous system disorders) | 12 (12) | 4 (4)
Abdominal Pain (Gastrointestinal disorders) | 5 (5) | 3 (3)
Acne (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 4 (4)
Earache/infection (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (7)
Nausea/Vomiting (Gastrointestinal disorders) | 6 (6) | 5 (5)
Cold Symptoms (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 10 (10)
Increased Heart Rate (Cardiac disorders) | 1 (1) | 2 (2)
Low Blood Pressure (Vascular disorders) | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Aches (General disorders) | 4 (4) | 8 (8)
Weight Gain/Loss (General disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes